CLINICAL TRIAL: NCT03544216
Title: Accommodative Relief for Uncomfortable Non-Presbyopes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Principal Investigator, Erin Rueff, Clinical Research Optometrist and PhD Candidate, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2016H0382-60058303
Record Dates: First submitted 2017-01-12; First posted 2018-06-01 (Actual); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Asthenopia
Keywords: Contact Lens; Multifocal; Accommodation; Presbyopia
MeSH Terms: conditions — Asthenopia; Presbyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Single Vision First (Experimental): Subjects in this group will receive the single vision spherical (Bausch + Lomb ULTRA®) lens for the first two weeks and be crossed over to the multifocal (Bausch + Lomb ULTRA® for Presbyopia) lens for the second two weeks.Therefore, this group will receive both study interventions.
  Interventions: Device: Multifocal Contact Lens; Device: Single Vision Contact Lens
- Multifocal first (Experimental): Subjects in this group will receive the multifocal (Bausch + Lomb ULTRA® for Presbyopia) lenses for the first two weeks and be crossed over to the single vision spherical (Bausch + Lomb ULTRA®) lens for the second two weeks. Therefore, this group will receive both study interventions.
  Interventions: Device: Multifocal Contact Lens; Device: Single Vision Contact Lens

INTERVENTIONS:
Device: Multifocal Contact Lens — The multifocal contact lens (Bausch + Lomb ULTRA® for Presbyopia) will be worn for two weeks
Device: Single Vision Contact Lens — The single vision contact lens (Bausch + Lomb ULTRA®) will be worn for two weeks

SUMMARY:
This study will determine how multifocal contact lens correction affects symptoms of discomfort and asthenopia in a group of myopic contact lens wearers in the non-presbyopic age range (ages 30-40 years).

DETAILED DESCRIPTION:
The purpose of this study is to determine how multifocal contact lenses affect contact lens comfort in non-presbyopic contact lens wearers. Current soft contact lens wearers who have symptoms of discomfort in their contact lenses will be recruited. Each subject (n = 84) will wear a single vision soft contact lens (Ultra single vision spherical lens) for two weeks and a low add power multifocal (Ultra for Presbyopia) for two weeks. Half of the subjects will wear the single vision lens first, and half of the subjects will wear the multifocal lens first. Initial lens group will be chosen randomly. Subjects will complete surveys that assess their vision and comfort which each lens, and ocular surface and accommodative/binocular vision status will be evaluated at the initial dispense and after wearing each lens for two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Visual acuity of 20/25 or better in both eyes with habitual contact lenses
* -0.75 D or more myopic in both eyes
* -0.75 D or less astigmatism in both eyes
* Current single vision contact lens wearer who does not require a reading aid
* CLDEQ-8 score of 12 or more points with habitual contact lenses
* No history of ocular surgery or medication
* Reports digital device use of at least 3 hours per day
* No significant signs of dry eye (grade 1 or less ocular surface staining, Schirmer score of 7 mm or more, and tear break up time of 7 seconds or more in bother eyes)
* No significant binocular vision disorders in both eyes (eso or exophoria of 4 prism diopters or less at distance and near, near point of convergence of 6 mm or less, no history of strabismus or patching)

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2018-05-06 (Actual); Study Completion 2018-05-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University College of Optometry, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Vision First: Subjects in this group will receive the single vision spherical (Bausch + Lomb ULTRA®) lens for the first two weeks and be crossed over to the multifocal (Bausch + Lomb ULTRA® for Presbyopia) lens for the second two weeks.
  Single Vision First, Multifocal Second: The single vision contact lens (Bausch + Lomb ULTRA®) will be worn for two weeks first, then the multifocal contact lens (Bausch + Lomb ULTRA® for Presbyopia) will be worn for two weeks
- Multifocal First: Subjects in this group will receive the multifocal (Bausch + Lomb ULTRA® for Presbyopia) lenses for the first two weeks and be crossed over to the single vision spherical (Bausch + Lomb ULTRA®) lens for the second two weeks.
  Multifocal First, Single Vision Second: The multifocal contact lens (Bausch + Lomb ULTRA® for Presbyopia) will be worn for two weeks first, then the single vision contact lens (Bausch + Lomb ULTRA®) will be worn for two weeks
Period: Overall Study
Arm/Group | Single Vision First | Multifocal First
Started | 42 | 42
Completed | 42 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Vision First | Multifocal First | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.4 (3.4) | 34.5 (3.1) | 34.4 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Data regarding gender of participants were not recorded for this study Population: Data regarding gender of participants were not recorded for this study.
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Data regarding race/ethnicity were not analyzed for this study. Population: Data regarding race/ethnicity were not analyzed for this study.
Contact Len Dry Eye Questionnaire-8 (CLDEQ-8) Score with Habitual Contact Lenses [Mean (Standard Deviation); unit: scores on a scale] — Min-Max range: 0-37 points Higher point values indicate more/worse symptoms
  scores on a scale | 19.0 (4.5) | 19.1 (5.0) | 19.0 (4.7)
Spherical Equivalent Refractive Error (Right Eye) [Mean (Standard Deviation); unit: diopters] | -4.2 (2.1) | -4.0 (2.0) | -4.1 (2.1)
Spherical Equivalent Refractive Error (Left Eye) [Mean (Standard Deviation); unit: diopters] | -4.2 (2.0) | -4.1 (2.0) | -4.2 (2.0)
Accommodative Lag with 2 Diopter Target [Mean (Standard Deviation); unit: diopters] — Accommodative Lag was measured with an autorefractor while the the subject was viewing a visual target at at 50 cm (2 diopter visual demand) and the single vision study lens. Accommdative lag is reported with the single vision lens only because the multifocal lens induces power changes that affect autorefractor measurements.
  diopters | 0.9 (0.5) | 0.8 (0.7) | 0.9 (0.6)
Accommodative Lag with 4 Diopter Target [Mean (Standard Deviation); unit: diopters] — Accommodative Lag was measured with an autorefractor while the the subject was viewing a visual target at at 25 cm (4 diopter visual demand) and the single vision study lens. Accommdative lag is reported with the single vision lens only because the multifocal lens induces power changes that affect autorefractor measurements.
  diopters | 1.3 (0.9) | 1.5 (0.7) | 1.4 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8) Score
Description: After wearing each lens type (single vision and multifocal) for 2 weeks, subjects will complete the CLDEQ-8, a survey that assesses symptoms of contact lens discomfort, to reports their symptoms of discomfort with each lens type. CLDEQ-8 scores with the multifocal will be compared to CLDEQ-8 scores of the single vision lens and the subjects' habitual contact lenses to determine if the multifocal improved comfort.
  Min-Max CLDEQ-8 range: 0-37 points Higher point values indicate more/worse symptoms
Time Frame: Baseline and after 2 weeks of contact lens wear with each study lens (single vision and multifocal)
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- CLDEQ-8 With Multifocal Contact Lens: Mean CLDEQ-8 score across both groups (single vision first and multifocal first)(n = 84) with the multifocal contact lens
- CLDEQ-8 With Single Vision Contact Lens: Mean CLDEQ-8 score across both groups treatment groups (single vision first and multifocal first)(n = 84) with the single vision contact lens
- CLDEQ-8 With Habitual Contact Lenses: Mean CLDEQ-8 score across both groups (single vision first and multifocal first)(n=84) at baseline with each subject's habitual contact lenses
Arm/Group | CLDEQ-8 With Multifocal Contact Lens | CLDEQ-8 With Single Vision Contact Lens | CLDEQ-8 With Habitual Contact Lenses
Number analyzed (Participants) | 84 | 84 | 84
scores on a scale | 14.3 (7.1) | 12.8 (6.6) | 19.0 (4.7)
Statistical Analysis 1: Comparison: CLDEQ-8 With Multifocal Contact Lens vs CLDEQ-8 With Single Vision Contact Lens vs CLDEQ-8 With Habitual Contact Lenses; Generalized linear models (controlling for repeated measures) of crossover analyses was run to compare mean CLDEQ-8 scores with habitual, multifocal, and single vision contact lenses (controlling for order); Test type: Other; p < 0.001, Generalized linear models — Results of post-hoc analyses comparing scores of each lens type to one another: Habitual lens and multifocal contact lens: p <0.001 Habitual lens and single vision lens: p <0.001 Multifocal lens and single vision lens: p = 0.08
Statistical Analysis 2: Comparison: CLDEQ-8 With Multifocal Contact Lens vs CLDEQ-8 With Single Vision Contact Lens; A generalized linear model was run to determine if there was an interaction between lens type (single vision or multifocal) and refractive error (continuous, mean binocular spherical equivalent); Test type: Other; p = 0.5, Generalized linear model — Analysis controlled for order, visit, and repeated measures
Statistical Analysis 3: Comparison: CLDEQ-8 With Multifocal Contact Lens vs CLDEQ-8 With Single Vision Contact Lens; A generalized linear model was run to determine if there was an interaction between magnitude in accommodative lag (measured in diopters with a 2 diopter visual target) and lens type (single vision or multifocal); Test type: Other; p = 0.7, Generalized linear model — Analysis controlled for order, visit, and repeated measures
Statistical Analysis 4: Comparison: CLDEQ-8 With Multifocal Contact Lens vs CLDEQ-8 With Single Vision Contact Lens; A generalized linear model was run to determine if there was an interaction between lens type (single vision or multifocal) and age (continuous, measured in self-reported years); Test type: Other; p = 0.3, Generalized linear model — Analysis controlled for order, visit, and repeated measures
Statistical Analysis 5: Comparison: CLDEQ-8 With Multifocal Contact Lens vs CLDEQ-8 With Single Vision Contact Lens; A generalized linear model was run to determine if there was an interaction between lens type (single vision or multifocal) and age (measured categorically as 30 to <35 years old and 35 to 40 years old, by self report); Test type: Other; p = 0.047, Generalized linear model — Analysis controlled for order, visit, and repeated measures; Post-Hoc Testing comparing CLDEQ-8 scores and the interaction between lens type and age group (denoted by lens type*age group) produced the following results: p = 0.01 for MF*<35 age group compared to Single Vision (SV)*<35 age group p = 0.07 for MF*<35 age group compared to MF*>35 age group p > 0.05 for MF*<35 age group compared to Single Vision (SV)*>35 age group p > 0.05 for SV*<35 age group compared to SV*>35 age group p >0.05 for SV*<35 age group compared to MF*>35 age group p > 0.05 for MF*>35 age group compared to SV*>25 age group

ADVERSE EVENTS:
Time Frame: Data from potential adverse events were collected for the duration of the study for each subject. From baseline to final visit, each subject participated in the study for approximately 4-6 weeks.
Groups:
- Single Vision Contact Lens: All subjects wore the single vision (Bausch + Lomb ULTRA®) lens for approximately 2 weeks during the study.
- Multifocal Contact Lens: All subjects wore the multifocal vision (Bausch + Lomb ULTRA® for Presbyopia) lens for approximately 2 weeks during the study.
Arm/Group | Single Vision Contact Lens | Multifocal Contact Lens
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/84
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/84
Other Adverse Events (participants affected / at risk) | 0/84 | 0/84

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT03544216/Prot_SAP_000.pdf